CLINICAL TRIAL: NCT05458375
Title: Vaginal Estradiol Use in Pessary Management: A Randomized Controlled Trial
Brief Title: Vaginal Estradiol Use in Pessary Care
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: There is a lack of potential study participants at our study site that would meet inclusion criteria, therefore, the study is not feasible and is being terminated.
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY004394
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-06

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Pessary Ulcer of Vagina; Vaginal Atrophy
Keywords: pessary; vaginal estradiol
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: The study design will be a randomized controlled trial involving patients seen in the Urogynecology clinic with pelvic organ prolapse or incontinence who were recently fit with a pessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (No Intervention): Participants will receive standard pessary care. Participation requires follow up visit 6 months from initial baseline visit. At this visit, participants are asked about vaginal bleeding, degree of bother due to vaginal discharge, and degree of pessary discomfort and a physical exam is performed.
- Estrogen Group (Experimental): Participants will receive standard pessary care, and those participants randomized to the experimental group will then be given a prescription for vaginal estradiol and instructed to apply it in the vagina nightly for two weeks and then twice weekly thereafter. Participation requires follow up visit 6 months from initial baseline visit. At this visit, participants are asked about vaginal bleeding, degree of bother due to vaginal discharge, and degree of pessary discomfort and a physical exam is performed.
  Interventions: Drug: Estradiol vaginal cream

INTERVENTIONS:
Drug: Estradiol vaginal cream — Insert pea-sized amount of vaginal estradiol cream into vagina nightly for first two weeks and then twice weekly thereafter.
  Other Names: Estrace; National Drug Code 0430-3754
  Arms: Estrogen Group

SUMMARY:
The primary outcome of this study compare the rate of pessary discontinuation at 6 months post-pessary fitting in women using vaginal estradiol versus those not using vaginal estradiol.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effects of vaginal estradiol cream on pessary care. All patients presenting to the University of South Florida Urogynecology clinic for pessary fitting for pelvic organ prolapse and/or urinary incontinence are screened as potential study participants. After being informed of risks and benefits of participations and consent is obtained, patients that have been successfully fitted for a pessary and agree to participate will be separated into two groups: the control group or treatment group. The treatment group will be provided with a prescription for vaginal estradiol cream. Vaginal estradiol cream is FDA approved and is the first line treatment for vaginal atrophy, also known as dryness. The study will be unblinded and randomized, neither the participant nor the study doctor will choose which group the will be participant will be placed in. The participant will have an equal chance of being given either treatment. The treatment group will be asked to apply vaginal estradiol cream nightly for two weeks and then twice weekly thereafter. All participants will have 2 study visits over a 6-month period which is standard for pessary care: a regular follow up pessary check visit two weeks after pessary fitting and second visit 6 months later. At these visits, questions regarding symptoms including vaginal bleeding, vaginal discharge, and discomfort with pessary will be assessed and a physical exam will be performed as is standard for all pessary users.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Postmenopausal status
* Recent pessary fitting
* Office-based and home-based pessary care

Exclusion Criteria:

* Women < 18 years old
* Women currently on hormone replacement therapy (pill, patch, pellet)
* Women currently using vaginal estradiol cream within the last 4 weeks
* Medical contraindications to vaginal estradiol including unevaluated vaginal bleeding
* Inability to apply vaginal estradiol cream
* Inability to provide informed consent
* Inability to comprehend written and/or spoken English or Spanish
* Inability to comply with study visit schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Pessary Discontinuation Rates | 6 Months Post-Pessary Fitting
  To compare the rate of pessary discontinuation at 6 months post-pessary fitting in estrogen group and no intervention group

SECONDARY OUTCOMES:
Phone calls/messages | 6 Months Post-Pessary Fitting
  To compare the number of phone calls/messages from patients to the office regarding pessary management symptoms in estrogen group and no intervention group
Unscheduled office visits | 6 Months Post-Pessary Fitting
  To compare the number of unscheduled office visits from patients in estrogen group and no intervention group
Vaginal Bleeding | Baseline Visit (Pessary Fitting), Final Visit (6 Months Post-Pessary Fitting)
  To compare the rates of vaginal bleeding from patients in estrogen group and no intervention group. As is standard in our practice, the pessary check visit includes an interview with the patient where specific self-reported symptoms are assessed. Participants will answer with self-reported "yes/no" during interview at the baseline study visit and at the final study visit.
Pessary Discomfort | Baseline Visit (Pessary Fitting), Final Visit (6 Months Post-Pessary Fitting)
  To compare the degrees of pessary discomfort using visual analogue scale measured in millimeters between patients in estrogen group and no intervention group. On this scale, the value 1 reflects no complaints of this side-effect and 10 reflects very severe complaints of this side-effect.
Vaginal Discharge | Baseline Visit (Pessary Fitting), Final Visit (6 Months Post-Pessary Fitting)
  To compare the degrees of bother of vaginal discharge using visual analogue scale measured in millimeters between patients in estrogen group and no intervention group. On this scale, the value 1 reflects no complaints of this side-effect and 10 reflects very severe complaints of this side-effect.
Urinary Tract Infection Rates | Final Visit (6 Months Post-Pessary Fitting)
  To compare the rates of urinary tract infections between patients in estrogen group and no intervention group. The diagnosis of urinary tract infection (UTI) is based on confirmatory testing, specifically with urine culture.
Vaginal Erosion Rates | Final Visit (6 Months Post-Pessary Fitting)
  To compare the rates of vaginal erosions between patients in estrogen group and no intervention group. Any vaginal erosions will be noted during the vaginal exam at the final visit, which is standard in our practice. Vaginal erosions are described using the following definitions: Type 0: No abnormalities; Type 1: Epithelial erythema; Type 2: Granulation tissue; Type 3: Epithelial break or erosion ≤ 1 cm; Type 4: Epithelial break or erosion > 1 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra N Garcia, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clemons JL, Aguilar VC, Tillinghast TA, Jackson ND, Myers DL. Risk factors associated with an unsuccessful pessary fitting trial in women with pelvic organ prolapse. Am J Obstet Gynecol. 2004 Feb;190(2):345-50. doi: 10.1016/j.ajog.2003.08.034. PMID 14981372
- [Background] Wolff B, Williams K, Winkler A, Lind L, Shalom D. Pessary types and discontinuation rates in patients with advanced pelvic organ prolapse. Int Urogynecol J. 2017 Jul;28(7):993-997. doi: 10.1007/s00192-016-3228-9. Epub 2016 Dec 10. PMID 27942793
- [Background] Dessie SG, Armstrong K, Modest AM, Hacker MR, Hota LS. Effect of vaginal estrogen on pessary use. Int Urogynecol J. 2016 Sep;27(9):1423-9. doi: 10.1007/s00192-016-3000-1. Epub 2016 Mar 18. PMID 26992727
- [Background] Bulchandani S, Toozs-Hobson P, Verghese T, Latthe P. Does vaginal estrogen treatment with support pessaries in vaginal prolapse reduce complications? Post Reprod Health. 2015 Dec;21(4):141-5. doi: 10.1177/2053369115614704. Epub 2015 Nov 3. PMID 26537626
- [Background] Propst K, Mellen C, O'Sullivan DM, Tulikangas PK. Timing of Office-Based Pessary Care: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jan;135(1):100-105. doi: 10.1097/AOG.0000000000003580. PMID 31809432
- [Background] Tontivuthikul P, Sanmee U, Wongtra-Ngan S, Pongnarisorn C. Effect of Local Estrogen Cream on Vaginal Health after Pessary Use for Prolapsed Pelvic Organ: A Randomized Controlled Trial. J Med Assoc Thai. 2016 Jul;99(7):757-63. PMID 29901374
- [Background] Cundiff GW, Weidner AC, Visco AG, Bump RC, Addison WA. A survey of pessary use by members of the American urogynecologic society. Obstet Gynecol. 2000 Jun;95(6 Pt 1):931-5. doi: 10.1016/s0029-7844(00)00788-2. PMID 10831995
- [Background] Lough K, Hagen S, McClurg D, Pollock A; JLA Pessary PSP Steering Group. Shared research priorities for pessary use in women with prolapse: results from a James Lind Alliance Priority Setting Partnership. BMJ Open. 2018 Apr 28;8(4):e021276. doi: 10.1136/bmjopen-2017-021276. PMID 29705767